CLINICAL TRIAL: NCT01910779
Title: Optimization of Initial Energy for Cardioversion of Atrial Fibrillation With Biphasic Shocks (OPTIMA Trial).
Brief Title: Optimization of Initial Energy for Cardioversion of Atrial Fibrillation With Biphasic Shocks
Acronym: OPTIMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Vittoria Hospital (Other)
Responsible Party: Principal Investigator, Massimo Imazio, MD, Maria Vittoria Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18/04/13
Record Dates: First submitted 2013-07-24; First posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Atrial Fibrillation; Cardioversion
Keywords: Atrial Fibrillation; Cardioversion; Biphasic Shock
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 100 joule arm (Active Comparator): 100 joule as first biphasic shock energy
  Interventions: Procedure: 100 joule as first biphasic shock energy
- 120 joule arm (Active Comparator): 120 joule as first biphasic shock energy
  Interventions: Procedure: 120 joule as first biphasic shock energy

INTERVENTIONS:
Procedure: 100 joule as first biphasic shock energy
  Arms: 100 joule arm
Procedure: 120 joule as first biphasic shock energy
  Arms: 120 joule arm

SUMMARY:
Use of higher energy doses (120-150 J) may not offer additional benefits and higher success rate compared with low to moderate initial energy (100-120 J) of biphasic shock for atrial fibrillation cardioversion. In this prospective open-label randomized trial consecutive patients with AF and candidate to AF electrical cardioversion will be randomized to receive 100J or 120 J as initial dose of biphasic shock. Patients will be also randomized in each group to anterolateral or postero-anteriore placement of defibrillator electrodes.

DETAILED DESCRIPTION:
Open-label randomized trial to assess the efficacy of alternative initial biphasic shocks (100 versus 120 J) for cardioversion of atrial fibrillation including alternative option for electrode placement (anterolateral or postero-anterior in each group).

ELIGIBILITY:
Inclusion Criteria:

* Adult (Age>18 years)
* Candidate to Cardioversion for recent onset, persistent atrial fibrillation (>48 hours but < 12 months)
* Informed Consent

Exclusion Criteria:

* Atrial Flutter or other arrythmias

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Electrical cardioversion success | Day 1

SECONDARY OUTCOMES:
Electrical cardioversion success | 3 months
Complications rate | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Imazio, MD, Principal Investigator — Cardiology Dpt. Maria Vittoria Hospital, Torino, Italy
Locations (1):
- Cardiology Dpt. Maria Vittoria Hospital, Torino, Torino, Italy